CLINICAL TRIAL: NCT02376101
Title: Minimal Occlusive Pressure With Cuffed ETT: the Effect of Size on Intracuff Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB14-00521
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Intracuff Pressure; ETT Size

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard ETT size (Active Comparator): Their tracheas will be intubated with an appropriately sized ETT using the standard formula. The cuff will be inflated to achieve a seal by the air-leak test when holding CPAP of 20 cmH2O and the intracuff pressure will be measured using a manometer.
  Interventions: Procedure: Surgery less than 60 minutes
- ETT one size smaller (Experimental): Their tracheas will be intubated with an ETT that is one size smaller (instead of a 5.0 ETT, we would use a 4.0 ETT). The cuff will be inflated to achieve a seal by the air-leak test when holding CPAP of 20 cmH2O and the intracuff pressure will be measured using a manometer.
  Interventions: Procedure: Surgery less than 60 minutes

INTERVENTIONS:
Procedure: Surgery less than 60 minutes

SUMMARY:
The purpose of this current study is to evaluate whether the size of the endotracheal tube (ETT) that is used impacts the intracuff pressure that occurs when the airway is sealed. If there is excessive pressure in the cuff of a smaller ETT when it is inflated, there may be inherent risks associated with the use of a cuffed endotracheal tube that is less than the appropriate size. The investigators believe that the size of the tube chosen has an impact on the characteristics of the inflated cuff and hence the intracuff pressure and the sealing pressure are variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intubation with an ETT for a surgical procedure.
* Children ages 4 to 8 years old.
* Surgical procedure lasting less than 60 minutes.

Exclusion Criteria:

* Patients undergoing a surgical procedure that is anticipated to last longer than 60 minutes.
* Patients that are known or anticipated to have a difficult airway.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Intracuff pressure | intraoperative
  Our goal is to measure the intracuff pressure that is achieved when the airway is sealed with an ETT based on the formula (ETT=(age/4)+3) and compare it to the intracuff pressure when the airway is sealed with an ETT that is 1 size smaller (4.0 mm instead of 5.0 mm).